CLINICAL TRIAL: NCT05687981
Title: The Analgesic Efficacy of Two Bupivacaine Concentrations for Combined Ilioinguinal and Iliohypogastric Nerve Block in Postherniorrhaphy Pain.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mariam Jamal Elkasass, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (IIIH) &(IINB) in pain control
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Hernia, Inguinal
Keywords: nerve block
MeSH Terms: conditions — Hernia, Inguinal | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients will receive 10 ml of 0.5% bupivacaine (Active Comparator): A 2mg dexamethasone will be added
  Interventions: Drug: Bupivacaine
- Patients will receive 10 ml of 0.25% bupivacaine (Active Comparator): A 2mg dexamethasone will be added
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine — the use of higher concentration of bupivacaine in ilioinguinal and iliohypogastric nerve block (IINB) might increase the efficacy of postoperative analgesia
  Arms: Patients will receive 10 ml of 0.5% bupivacaine
Drug: Dexamethasone — 2 mg dexamethasone
  Arms: Patients will receive 10 ml of 0.25% bupivacaine

SUMMARY:
The present study will be undertaken to compare the postoperative analgesic effect of 0.25% bupivacaine and 0.5% bupivacaine for unilateral ilioinguinal and Iliohypogastric nerve block after open inguinal hernia repair.

Primary outcome:

The time to first request for rescue analgesia.

Secondary outcome:

1. The post-operative pain in the form of NRS scores at rest & during movement at 0, 2, 4, 8, 12, 18 and 24 hours post-procedure.
2. The total 24 hour opioid consumption.
3. The incidence of complication related to nerve block (urinary retention, hematoma, hypotension and arrhythmia).
4. Patient satisfaction

DETAILED DESCRIPTION:
Postoperative pain is a common complication that may cause a neuroendocrine stress response, which is characterized by increased release of catabolic and immunosuppressive pituitary hormones and activation of the sympathetic nervous system. Excessive postoperative pain and the physiological stress response can influence postoperative outcomes, length of hospital stay and overall costs of hospital care Inguinal herniorrhaphy is a common outpatient surgical procedure with approximately 20 million operations performed worldwide annually.

Patients undergoing this procedure often experience moderate-to-severe pain, which can hinder post anesthesia care unit (PACU) discharge. While pain can be treated with opioid therapy, the literature supports that opioids may cause postoperative nausea, vomiting, hypoxia, and urinary retention. In contrast, analgesia provided by regional block has been shown to decrease the previous complications.

There is an ongoing interest in developing regional anesthetic techniques that may reduce or eliminate the use of opioid analgesics after minor surgical procedures such as hernia repair.

Regional analgesia has found wide acceptance both by the patients and their treating physicians, and therefore, it is now an important part of multimodal analgesia techniques. Ilioinguinal/iliohypogastric nerve block(IINB),transversus abdominis plane (TAP) block, paravertebral and rectus sheath, have all been used for providing analgesia following abdominal surgeries .

The combined ilioinguinal and iliohypogastric nerve block (IINB) is a commonly used technique for blockade of the ilioinguinal/iliohypogastric (IIIH) nerves and has been shown to decrease pain after OIH as well as reduce opioid requirements.

Bupivacaine belongs to the amide family, and its structure is similar to that of lidocaine. Bupivacaine is a potent agent capable of producing prolonged anesthesia. Its long duration of action plus its tendency to provide more sensory than motor block has made it a popular drug for providing prolonged analgesia during the postoperative period.

We assume that the use of higher concentration of bupivacaine in ilioinguinal and iliohypogastric nerve block (IINB) might increase the efficacy of post-operative analgesia and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 21 and 60 years age with the American Society of Anesthesiologists' status I or II scheduled for elective primary open inguinal hernia repair

Exclusion Criteria:

1. Patient refusal.
2. Body mass index (BMI) >40 kg m2.
3. The presence of skin infection at the injection site.
4. Allergy to local anesthetic drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
The time to first request for rescue analgesia. | 24 hours
  if score is ≥ 3 analgesia needed

SECONDARY OUTCOMES:
The post-operative pain in the form of NRS. | at 0, 2, 4, 8, 12, 18 and 24 hours post-procedure.
The total 24 hour opioid consumption | 24 hours
The incidence of complication related to nerve block | 48 hours
  urinary retention, hematoma, hypotension and arrhythmia
Patient satisfaction | 48 hours
  in the form of 4 point satisfaction questionnaire: where 1 would be satisfied, 2=neutral, 3=dissatisfied, and 4=extremely dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Abduallah, Study Director — Tanta University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bugedo GJ, Carcamo CR, Mertens RA, Dagnino JA, Munoz HR. Preoperative percutaneous ilioinguinal and iliohypogastric nerve block with 0.5% bupivacaine for post-herniorrhaphy pain management in adults. Reg Anesth. 1990 May-Jun;15(3):130-3. PMID 2265166
- [Background] Kamal K, Jain P, Bansal T, Ahlawat G. A comparative study to evaluate ultrasound-guided transversus abdominis plane block versus ilioinguinal iliohypogastric nerve block for post-operative analgesia in adult patients undergoing inguinal hernia repair. Indian J Anaesth. 2018 Apr;62(4):292-297. doi: 10.4103/ija.IJA_548_17. PMID 29720755